CLINICAL TRIAL: NCT02213133
Title: A Phase 2, Open-Label Study of the Safety and Efficacy of the Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Advanced Squamous Cell Carcinoma of the Head and Neck, Lung, or Esophagus
Brief Title: Selinexor Treatment of Advanced Relapsed/Refractory Squamous Cell Carcinomas
Acronym: STARRS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges and availability of other options for lung cancer patients. The termination is not a consequence of any safety concern.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-006
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: Squamous; SCC; Carcinoma; KPT-330; SINE; Selinexor; Karyopharm; Karyopharm Therapeutics; Lung; Head; Neck; Esophageal
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Head and Neck-SCC (Experimental): Participants with advanced squamous cell carcinoma (SCC) of head and neck, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 milligram (mg) selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets less than [<] 100*10^9 per litre [/L]), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
  Interventions: Drug: Selinexor (KPT-330)
- Cohort 2: Lungs-SCC (Experimental): Participants with advanced SCC of lungs, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 mg selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets <100*10^9/L), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
  Interventions: Drug: Selinexor (KPT-330)
- Cohort 3: Esophagus-SCC (Experimental): Participants with advanced SCC of esophagus, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 mg selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets <100*10^9/L), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
  Interventions: Drug: Selinexor (KPT-330)

INTERVENTIONS:
Drug: Selinexor (KPT-330) — Oral tablet or suspension at 60, 80, 100 or 120 mg per patient-specific body surface area category. Dosing will occur twice weekly in 28-days cycle.
  Other Names: KPT-330

SUMMARY:
Open-label, multi-center, single-arm, Phase 2 study of oral selinexor in patients with SCC of the head and neck (HN-SCC; Cohort 1), lung (L-SCC; Cohort 2), or esophagus (E-SCC; Cohort 3) who have relapsed or have metastasis following chemotherapy.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm Phase 2 study of the SINE selinexor given orally to patients diagnosed with advanced SCC of the head and neck, lung, or esophagus who have experienced relapse and/or metastasis following multiple prior chemotherapy treatments (<2 lines of therapy).

Patients will receive fixed doses of selinexor tablets twice weekly in 28-day cycles. Patients may continue from one cycle to the next without interruption as along as all criteria are met and no reason for discontinuation occurs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* confirmed SCC of the head and neck, lung, or esophagus
* 1 to 2 prior therapies
* measurable disease at screening and documented progression within the past 6 weeks

Exclusion Criteria:

* patients requiring total parenteral nutrition
* unstable cardiovascular function
* substantially impaired gastrointestinal function
* Symptomatic brain metastases
* another malignancy within 3 years except adequately treated in situ carcinoma of any type, basal or non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute / Harvard University, Boston, Massachusetts
  - Metrowest Medical Center, Framingham, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine / Washington University in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Herbert Irving Comprehensive Cancer Center / Columbia University, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center / Vanderbilt University, Nashville, Tennessee
  - Mary Crowley Cancer Research Center / Texas Oncology, Dallas, Texas
  - University of Washington, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in United States and 1 site in Canada between 22 September 2014 and 10 December 2015.
Pre-assignment Details: A total of 45 participants were enrolled and randomized.
Groups:
- Cohort 1: Head and Neck-SCC: Participants with advanced squamous cell carcinoma (SCC) of head and neck, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 milligrams (mg) selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets less than [<] 100*10^9 per litre [/L]), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
Period: Overall Study
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Cohort 3: Esophagus-SCC
Started (Enrolled) | 37 | 5 | 3
Treated | 33 | 4 | 1
Completed | 0 | 0 | 0
Not Completed | 37 | 5 | 3
Not completed — Participant discontinued study therapy | 2 | 0 | 0
Not completed — Participant withdrew informed consent | 2 | 1 | 2
Not completed — Disease progression | 11 | 2 | 0
Not completed — Adverse Event (AE) | 1 | 0 | 0
Not completed — Death | 16 | 2 | 1
Not completed — Other | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population (mITT) population included all participants who had received at least one dose of study drug and had at least one post baseline efficacy assessment were included if discontinuation was due to disease progression, study drug related toxicity, or death.
Groups:
- Cohort 1: Head and Neck-SCC: Participants with advanced SCC of head and neck, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 mg selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets <100*10^9/L), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Cohort 3: Esophagus-SCC | Total
Number analyzed (Participants) | 33 | 4 | 1 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.05) | 66.3 (6.34) | 51.0 (NA) — This arm reports single participant data, hence no data was analyzed for standard deviation for the specified arm. | 59.1 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 30 | 3 | 1 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 1 | 0 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 0 | 0 | 0 | 0
  Race: White | 30 | 4 | 1 | 35
  Race: Other-unspecified | 1 | 0 | 0 | 1
  Race: Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Control Rate (DCR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: DCR was defined as the best overall response of complete response (CR), partial response (PR), or stable disease (SD). CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Participant response was evaluated by physical examinations and computed tomography (CT)/Magnetic Resonance Imaging (MRI) (or optional positron emission tomography [PET]/CT) and assessed by RECIST 1.1 criteria.
Time Frame: up to 14.6 months
Population: Analysis performed on mITT population that included all participants who received at least 1 dose of study drug, and had at least 1 post baseline efficacy assessment. Participants who discontinued prior to first post baseline efficacy assessment were included if discontinuation was due to disease progression, study drug related toxicity, or death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Cohort 3: Esophagus-SCC
Number analyzed (Participants) | 33 | 4 | 1
percentage of participants | 21.2 [10.7 to 37.8] | 0.0 [0.0 to 49.0] | 0.0 [0.0 to 79.3]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any unfavorable sign and unintended sign (including abnormal laboratory finding), symptom, or disease temporarily associated with the use of the study drug, whether or not related to study drug. An SAE was defined as any untoward medical occurrence that occurs at any dose (including after informed consent was signed and prior to dosing) that resulted in death, was life-threatening (participant was at immediate risk of death from event), required in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect, and important medical events. A TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after first dose of treatment through 30 days following last dose of study treatment, or any event considered drug-related by investigator through end of study.
Time Frame: From the first administration of study drug up to 30 days follow-up (up to 14.6 months)
Population: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Lungs-SCC; Cohort 3: Esophagus-SCC: Participants with advanced SCC of esophagus, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 mg selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets <100*10^9/L), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Cohort 3: Esophagus-SCC
Number analyzed (Participants) | 37 | 5 | 3
Participants
  Participants with TEAEs | 37 | 5 | 3
  Participants with SAEs | 18 | 2 | 3

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events by Severity: Clinical Terminology Categories for Adverse Events (CTCAE) Grading Scale
Description: AE:Any unfavorable sign and unintended sign,symptom, or disease temporarily associated with use of study drug, whether or not related to it. SAE:Any untoward medical occurrence that occurs at any dose (after informed consent was signed, prior dosing) that resulted in death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, and important medical events. TEAE:Any AE with onset or worsening of existing condition on or after first dose through 30 days following last dose of study drug, or any event considered drug-related by investigator through end of study. Severity(Grades 1 to 5) of each AE was categorized as either mild=1(transient,does not interfere with daily activities), moderate=2(low level of inconvenience or concern,interfere with daily activities), severe=3(interrupt usual daily activities), life threatening=4 or fatal=5, higher grade reported worst outcome.
Time Frame: From the first administration of study drug up to 30 days follow-up (up to 14.6 months)
Population: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Cohort 3: Esophagus-SCC
Number analyzed (Participants) | 37 | 5 | 3
Participants
  Mild (Grade 1) | 3 | 0 | 0
  Moderate (Grade 2) | 9 | 1 | 0
  Severe (Grade 3) | 21 | 4 | 3
  Life Threatening (Grade 4) | 3 | 0 | 0
  Fatal (Grade 5) | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first administration of study drug up to 30 days after participant's last visit (up to 14.6 months)
Description: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Groups:
- Esophagus-SCC: Participants with advanced SCC of esophagus, who had relapsed or had metastasis following chemotherapy, received a fixed dose of 60 mg selinexor oral tablets twice weekly on Days 1 and 3 of a 28-day cycle (8 doses in 4 weeks) until disease progression or development of unacceptable toxicities. After completion of Cycle 2, for participants with absence of any grade 2 toxicity and thrombocytopenia (platelets <100*10^9/L), dose may be increased to 80 mg selinexor oral tablets twice weekly as assessed by investigator in a 28-day cycle until disease progression or development of unacceptable toxicities.
Arm/Group | Cohort 1: Head and Neck-SCC | Cohort 2: Lungs-SCC | Esophagus-SCC
All-Cause Mortality (participants affected / at risk) | 16/37 | 2/5 | 1/3
Serious Adverse Events (participants affected / at risk) | 18/37 | 2/5 | 3/3
Other Adverse Events (participants affected / at risk) | 35/37 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Head and Neck-SCC (N=37) | Cohort 2: Lungs-SCC (N=5) | Esophagus-SCC (N=3)
Pneumonia (Infections and infestations) | 5 | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 2
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tracheal Obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Head and Neck-SCC (N=37) | Cohort 2: Lungs-SCC (N=5) | Esophagus-SCC (N=3)
Nausea (Gastrointestinal disorders) | 25 | 4 | 0
Vomiting (Gastrointestinal disorders) | 13 | 2 | 0
Constipation (Gastrointestinal disorders) | 10 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 21 | 4 | 1
Pyrexia (General disorders) | 3 | 0 | 2
Asthenia (General disorders) | 3 | 1 | 0
Face Oedema (General disorders) | 4 | 0 | 0
Chills (General disorders) | 3 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 12 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Weight Decreased (Investigations) | 6 | 1 | 0
Platelet Count Decreased (Investigations) | 3 | 1 | 1
Blood Creatinine Increased (Investigations) | 2 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Confusional State (Psychiatric disorders) | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Lung Infection (Infections and infestations) | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Vision Blurred (Eye disorders) | 6 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to enrollment challenges and availability of other options for lung cancer participants. The termination was not a consequence of any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes